CLINICAL TRIAL: NCT06162559
Title: Neoadjuvant Trastuzumab, Pertuzumab and Tucatinib Without Chemotherapy in HER2-positive Breast Cancer: the TRAIN-4 Study
Acronym: TRAIN-4
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: The Netherlands Cancer Institute (Other)
Collaborators: Seagen Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N21TRV
Record Dates: First submitted 2023-11-29; First posted 2023-12-08 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: Breast Cancer
Keywords: neoadjuvant; HER2 positive; tucatinib; Breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — tucatinib; Trastuzumab; pertuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tucatinib + trastuzumab + pertuzumab (Experimental): All patients receive neoadjuvant treatment consisting of trastuzumab, pertuzumab and tucatinib. Patients with hormone receptor positive disease receive concurrent endocrine therapy with an aromatase-inhibitor. Premenopausal women are concurrently treated with a LHRH-agonist. In case of functional tumor volume decrease of at least 65% (responders) after the first three cycles, patients continue treatment for six more cycles of the chemotherapy-free regimen. If tumor response is <65% (non-responders), patients will switch to receive six cycles paclitaxel, carboplatin, trastuzumab and pertuzumab. This is considered non-investigational treatment.
  Interventions: Drug: Tucatinib; Drug: Trastuzumab; Drug: Pertuzumab

INTERVENTIONS:
Drug: Tucatinib — Tucatinib 300mg is taken orally twice daily
  Other Names: Tukysa
Drug: Trastuzumab — Trastuzumab 6mg/kg is administered intravenously on day 1 (loading dose 8mg/kg) or subcutaneously 600mg on day 1 of each cycle
  Other Names: Herceptin
Drug: Pertuzumab — Pertuzumab 420mg is administered intravenously on day 1 (loading dose 840mg) or subcutaneously 600mg/kg (loading dose 1200mg) on day 1 of each cycle
  Other Names: Perjeta

SUMMARY:
This is a single-center, phase 1b study evaluating the safety and feasibility of a neoadjuvant treatment with tucatinib, trastuzumab and pertuzumab in stage II-IIIA HER2-positive breast cancer.

DETAILED DESCRIPTION:
High pathological complete response (pCR)-rates are seen using different neoadjuvant chemotherapy schedules with trastuzumab and pertuzumab in HER2-positive stage II - III breast cancer patients. However, a subset of patients with stage II-III HER2-positive breast cancer can be treated with HER2-blockade alone. These patients can potentially be totally spared from chemotherapy-associated toxicity. The proportion of patients whom can successfully be treated without chemotherapy could potentially be increased by selecting great responders using DCE-MRI and by adding tucatinib to trastuzumab and pertuzumab alone. The aim of this study is to evaluate the safety and efficacy of neoadjuvant treatment with tucatinib, trastuzumab and pertuzumab.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent
2. Histologically confirmed primary invasive breast cancer
3. Stage II - IIIA primary breast cancer according to TNM-staging (8th edition, AJCC); (largest tumor diameter on DCE-MRI ≥ 2cm (cT2-3) and/or cN1-2 confirmed with FNA or histology)
4. HER2 overexpression defined as circumferential membrane staining that is complete, intense and in >10% of invasive tumor cells (IHC 3+) on pre-treatment biopsy
5. Known estrogen- and progesterone-receptor expression of the invasive tumor

   a. ER-negative or PR-negative is defined as <10% of invasive tumor cell nuclei are immunoreactive in the presence of evidence that the sample can express ER and/or PR
6. WHO performance status 0-1
7. Age ≥ 18 years
8. LVEF ≥50% measured by echocardiography or MUGA
9. Eligible for neoadjuvant treatment
10. Laboratory requirements within 21 days prior to enrollment:

    1. Adequate bone marrow function (ANC ≥1.5 x 109/l, platelets ≥100 x 109/l);
    2. Adequate hepatic function (ALAT, ASAT and bilirubin ≤2.5 times upper limit of normal). Subjects with Gilbert's syndrome may have a total bilirubin ≥2.5 × the ULN range, if no evidence of biliary obstruction exists.
    3. Adequate renal function: creatinine clearance >50 ml/min estimated using the Cockcroft-Gault equation or MDRD equation, or based on a 24-hour urine collection measurement.

Exclusion Criteria:

1. Current pregnancy or breastfeeding
2. Current or previous other malignancy unless treated without systemic therapy and more than five years ago
3. Psychological, familial, sociological, or geographical condition potentially hampering compliance with the study protocol and follow-up schedule
4. Use of a strong CYP3A4 or CYP2C8 inhibitor within five half-lives of the inhibitor, or used a strong CYP3A4 or CYP2C8 inducer within five days prior to first dose of study treatment
5. Known chronic liver disease
6. History of inflammatory bowel disease or bowel resection
7. Contraindications for MRI
8. Inflammatory breast cancer, cT4 and/or cN3 tumors
9. Occult breast cancer (cT0)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-12-18 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2036-05 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of adverse events | an average of 8 months
  Number of patients with adverse events and severity of adverse events (all grades; CTCAE v5.0) until 30 days after last study treatment administration

SECONDARY OUTCOMES:
Incidence of serious adverse events | an average of 8 months
  Number of patients with serious adverse events until 30 days after last study treatment administration
Incidence of disease progression | an average of 8 months
  Number of patients with progressive disease during neoadjuvant treatment. Progressive disease is defined as 20% increase in ∆FTV or >20% increase measured in the longest diameter on DCE-MRI or unequivocal new lesions on (18)F-FDG PET
Incidence of dose reductions and treatment discontinuations | an average of 8 months
  Number of patients with dose reductions and treatment discontinuations
Radiologic complete response | an average of 8 months
  Number of patients with a radiologic complete response defined as the absence of pathologic enhancement on contrast enhanced MRI breast
Pathological complete response | an average of 8 months
  Number of patients with a pathological complete response (ypT0/is N0) at surgery in patients treated without chemotherapy, and overall
Residual Cancer Burden | an average of 8 months
  Residual Cancer burden (RCB, 0-III) at surgery in patients treated without chemotherapy, and overall
Event-free survival | 3, 5, 10 years
  Number of patients without progression or disease recurrence, second primary or death at 3, 5 and 10 years after registration
Overall survival | 3, 5, 10 years
  Number of patients alive at 3, 5 and 10 years after registration

CONTACTS AND LOCATIONS:
Locations (1):
- Netherlands Cancer Institute, Amsterdam, Netherlands